CLINICAL TRIAL: NCT04397549
Title: Evaluating the Effectiveness of Cervical Erector Spinae Block for Shoulder Surgery
Brief Title: Cervical Erector Spinae Block for Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konya Necmettin Erbakan Üniversitesi (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Alper Kilicaslan, MD, Assoc.Professor, Konya Necmettin Erbakan Üniversitesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ATA-173
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Pain; Shoulder Surgery
Keywords: cervical erector spinae plane block; postoperative pain; Shoulder Surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will randomized into two groups cervical ESP and control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Block group (Active Comparator): Cervical Erector Spinae Plane Block administered group
  Interventions: Other: Cervical erector spinae plane block; Device: Intravenous morphine patient controlled analgesia device
- Control group (Sham Comparator): Control group
  Interventions: Device: Intravenous morphine patient controlled analgesia device

INTERVENTIONS:
Other: Cervical erector spinae plane block — Cervical erector spinae plane block will be administered before the surgery
  Arms: Block group
Device: Intravenous morphine patient controlled analgesia device — 24 hour morphine consumption will be recorded

SUMMARY:
Arthroscopic shoulder surgery is often associated with moderate to severe postoperative pain that may interfere with patients' early mobilization, recovery and quality of life.

In addition, by using an effective analgesic technique, a patient may experience less nausea, vomiting and drowsiness after surgery that are associated with the use of opioids to manage postoperative pain. Erector spinae plane block (ESPB) has been used in many different indications for acute pain treatment at different thoracic and lumbar levels. Recently, staining the roots of the brachial plexus has been reported in a cadaveric study of the cervical ESPB (1).

However, there are only few case reports related to efficiency and safety of this newly defined cervical ESPB technique (2) .

The primary objective of this randomized controlled is investigate the post-operative analgesic effectiveness of ultrasound guided single-shot cervical ESPB for patients undergoing arthroscopic shoulder surgery in comparison to those receiving conventional parentheral opioid analgesia alone.

Secondary objective is testing the safety of this newly defined block in terms of incidence of complications.

DETAILED DESCRIPTION:
60 patients will be enrolled to in this study between June 2020 - October 2020. All patient will be randomly selected who will be operated for shoulder surgery. Age, weight, ASA score, body mass index, additional dissease status will be recorded. The patients will be divided in two groups. One group will have cervical ESPB before the operation and the second group will be treated with multimodal analgesia techniques and both groups will receive patient controlled analgesia.

Both groups will receive identical anaethesia protocols. Perioperative analgesia protocols will provide acetaminophen 1 gr and the same dose will be repeated in every 6 hours regardless of the pain scores. In postoperative period, the pain scores of the patients will be recorded according to the numeric rating scale (NRS) in every three hours. If pain score raises over 3/10 on NRS the patient will receive tramadol 100mg as rescue analgesia. In case of persisting pain first, meperidine 50 mg will be applied and other multimodal analgesic drugs will be added to protocol. At the end of the study 24 hours total opioid usage of patients, pain scores and side effects will statistically be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 18 -65 years of agge
* ASA I-II
* Undergoing elective shoulder surgery

Exclusion Criteria:

* infection of the skin at the site of needle puncture area
* patients with known allergies to any of the study drugs
* coagulopathy
* recent use of analgesic drugs
* obesity (body mass index >35 kg/m2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-15 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | 24 hour postoperatively
  All patients will be provided with IV morphine PCA and morphine consumption after 24 hour postoperatively will be recorded.

SECONDARY OUTCOMES:
Numering Rating Scale scores for pain | 24 hour
  Numeric Rating Scale (NRS) for pain will be used. The Numeric Rating Scale (NRS-11) is an 11- point scale for patient self-reporting of pain. It is for adults and children 10 years old or older. 0 means no pain and 10 means most imaginable pain
Postoperative nausea and vomiting | 24 hour
  Incidence of postoperative nausea and vomiting will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Alper Kilicaslan, MD, Assoc.Prof, Principal Investigator — Necmettin Erbakan University Meram Medical Faculty; İlker İnce, MD, Assoc.Prof, Principal Investigator — Ataturk University Medical Faculty
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hamadnalla H, Elsharkawy H, Shimada T, Maheshwari K, Esa WAS, Tsui BCH. Cervical erector spinae plane block catheter for shoulder disarticulation surgery. Can J Anaesth. 2019 Sep;66(9):1129-1131. doi: 10.1007/s12630-019-01421-9. Epub 2019 Jun 3. No abstract available. PMID 31161549
- [Result] Elsharkawy H, Ince I, Hamadnalla H, Drake RL, Tsui BCH. Cervical erector spinae plane block: a cadaver study. Reg Anesth Pain Med. 2020 Jul;45(7):552-556. doi: 10.1136/rapm-2019-101154. Epub 2020 Apr 21. PMID 32321860